CLINICAL TRIAL: NCT01761604
Title: The Use of Tx360™ Nasal Applicator for Sphenopalatine Ganglion Block in the Treatment of Trigeminal Neuralgia
Brief Title: A Nasal Applicator for the Treatment of Trigeminal Neuralgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chicago Anesthesia Pain Specialists (Other)
Responsible Party: Principal Investigator, Kenneth D Candido, Chairman of the Anesthesia Department at Advocate Illinois Masonic Medical Center, Chicago Anesthesia Pain Specialists
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Advocate-IRB-5241
Record Dates: First submitted 2013-01-02; First posted 2013-01-07 (Estimated); Last update posted 2017-09-14 (Actual); Status verified 2017-09

CONDITIONS: Trigeminal Neuralgia
MeSH Terms: conditions — Trigeminal Neuralgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nasal ganglion block for TN (Other): Sphenopalatine ganglion block using the Tx360™ device
  Interventions: Device: Nasal ganglion block for TN

INTERVENTIONS:
Device: Nasal ganglion block for TN

SUMMARY:
The pain from Trigeminal Neuralgia (TN) imposes a substantial burden on patients in daily function and reduces quality of life. The sphenopalatine ganglion, located in the posterior part of the middle nasal turbinate, is involved in the pain associated to TN, by blocking the sphenopalatine ganglion relieves patients from the symptoms. However, methods currently in use to accomplish this are either cumbersome for the patient or invasive regarding the puncture of structures.

The purpose of this study is to evaluate the efficacy of Tx360™, a new nasal applicator device, in the treatment of TN. A local anesthetic will be delivered on the ganglion area. We are expecting that this new device will provide at least the same pain relief as the previously described approaches. However, this nasal applicator is intended to be an easy and non invasive method for office use.

DETAILED DESCRIPTION:
The pain from Trigeminal Neuralgia (TN) imposes a substantial burden on patients in daily function and reduces quality of life. Pain severity correlates with reduced measures of daily functioning, and overall health status.

The sphenopalatine ganglion, located in the posterior part of the middle nasal turbinate, is involved in the pain associated to TN, by blocking the sphenopalatine ganglion relieves patients from the symptoms. However, methods currently in use to accomplish this are either cumbersome for the patient or invasive regarding the puncture of structures.

The purpose of this study is to evaluate the efficacy of Tx360™, a new nasal applicator device, in the treatment of TN. The Tx360™ is a single use nasal applicator that can reach the sphenopalatine ganglion area. It is designed to dispense medications through a flexible canula.

The patients with TN will receive a 0.5 mL spray of local anesthetic on the ganglion area, and measure the change in pain intensity and quality of life.

We are expecting that this new device will provide at least the same pain relief as the previously described approaches. However, this nasal applicator is intended to be an easy and non invasive method for office use.

ELIGIBILITY:
Inclusion Criteria:

* 18- 80 years old
* Trigeminal Neuralgia

Exclusion Criteria:

* Nasal septal deformity such as: cleft lip and palate, choanal atresia
* Septal perforation
* Recent nasal/midface trauma (< 3 months)
* Bleeding disorder such as Von Willebrand's disease or hemophilia
* Severe respiratory distress
* Neoplasm such as the following: Angiofibroma, sinus Tumors, Granuloma
* Congestion has been present more than 10 days, fever (define as temperature≥ 100.4 F)
* Current cocaine user
* Skin around and inside the nasal passage is dry, cracked, oozing, or bleeding
* Allergy to marcaine
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-12; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Pain intensity numeric rating scale | Before procedure and after procedure
  Change in pain intensity before procedure, baseline. And after procedure 15 minutes, 30 minutes, day 1, 7, 14, 21, and 28.

SECONDARY OUTCOMES:
Patient's global impression of change | After procedure
  Before procedure, baseline. And after procedure 30 minutes, day 1, 7, 14, 21, and 28.

OTHER OUTCOMES:
Modified Brief Pain inventory (short form) | Before procedure and after procedure
  Before procedure, baseline. And after procedure day 1, 7, 14, 21, and 28.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth D Candido, M.D., Principal Investigator — Chicago Anesthesia Pain Specialists
Locations (1):
- Chicago Anesthesia Pain Specialists, Chicago, Illinois, United States